CLINICAL TRIAL: NCT02616939
Title: Clinical In-hospital Evaluation of the Usefulness of a New Multi-detector Computed Tomography Scanner From Arineta Ltd
Acronym: Arineta
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: Arineta Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CMC-14-0127-CTIL
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: Multidetector computed tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with suspected cardiac disease: Patients eligible for cardiac CT will be included with a focus on symptomatic patients with low-intermediate risk for obstructive coronary artery disease.
  Patients will undergo Cardiac CT scanning (with the SpotLight CT).
  Interventions: Other: Cardiac CT scanning (with the SpotLight CT)

INTERVENTIONS:
Other: Cardiac CT scanning (with the SpotLight CT) — Cardiac CT scanning

SUMMARY:
Clinical evaluation of a new cardiovascular oriented CT scanner from Arineta Ltd.

DETAILED DESCRIPTION:
The study will evaluate a new twin source relatively compact CT scanner with advanced technology which is optimized for cardiovascular imaging. Eligible patients with a clinical indication will undergo coronary or cardiac CT scans using the new SpotLight CT from Arineta Ltd. Image quality and usefulness of the new system will then be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic patients with a clinical indication for cardiac CT
2. Patients with a clinical indication for CT
3. Estimated GFR > 60 mL/min

Exclusion Criteria:

1. No clinical indication for CT scanning
2. Contra-indication for CT scanning or for IV contrast administration
3. Pregnancy
4. Inability to give an informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical indication for cardiac CT
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Image quality (subjective) of the new SpotLight CT scanner from Arineta Ltd. | 2 years
  Subjective (4 grade scale) image quality assessment of coronary arteries. unassessable studies and unassessable coronary segments will be reported.
Image quality (objective) of the new SpotLight CT scanner from Arineta Ltd. | 2 years
  Image contrast, image noise, signal to noise ratio and contrast to noise ratio. Those numerical values will be reported to allow comparisons with values previously reported with other CT scanners.

SECONDARY OUTCOMES:
Diagnostic accuracy of the new SpotLight CT scanner from Arineta Ltd. | 2 years
  Performance characteristics of the new CT scanner for diagnosing obstructive coronary artery disease as compared to other reference standards such as invasive coronary angiography.
The effect of cardiac CT results (with SpotLight CT) on patients triage | 5 years
  The effect of cardiac CT results on patients diagnosis and therfore hospitalization or discharge decisions
The predictive value of cardiac CT results (with SpotLight CT) for patients outcome | 5 years
  Predictive value of cardiac CT results for adverse outcomes (death/myocardial infarction/revascularization).

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Rubinshtein, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No